CLINICAL TRIAL: NCT03119883
Title: Dysregulation of Glutamine Utilization in the Pathogenesis of Multiple Myeloma
Brief Title: Dysregulation of Glutamine Activity in the Pathogenesis of Multiple Myeloma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 17-003133; NCI-2021-02642 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); K23CA218742 (NIH)
Record Dates: First submitted 2017-04-12; First posted 2017-04-19 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Monoclonal Gammopathy of Undetermined Significance; Plasma Cell Myeloma
MeSH Terms: conditions — Monoclonal Gammopathy of Undetermined Significance; Multiple Myeloma | interventions — Specimen Handling; Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (biospecimen collection) (Experimental): EX-VIVO: After an overnight fast of 6 hours, patients undergo collection of bone marrow aspirate samples.
  Interventions: Procedure: Biospecimen Collection
- Group II (biospecimen collection, glutamine, glucose) (Experimental): IN VIVO: After an overnight fast of 6 hours, patients receive 13-carbon labeled glutamine or 13-carbon-labeled glucose IV over 90 minutes. Patients also undergo collection of blood and bone marrow aspirate samples.
  Interventions: Other: 5-Carbon C 13-labeled Glutamine; Procedure: Biospecimen Collection; Other: Uniformly-labeled [13C]glucose

INTERVENTIONS:
Other: 5-Carbon C 13-labeled Glutamine — Given IV
  Other Names: 5-13C-Glutamine; [5-13C]-glutamine; GLUTAMINE 5-C-13
  Arms: Group II (biospecimen collection, glutamine, glucose)
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
  Arms: Group II (biospecimen collection, glutamine, glucose)
Procedure: Biospecimen Collection — Undergo collection of bone marrow aspirate samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Uniformly-labeled [13C]glucose — Given IV
  Other Names: [U-13C] Glucose; U-13C-Glucose
  Arms: Group II (biospecimen collection, glutamine, glucose)

SUMMARY:
This clinical trial studies the utilization of glutamine by the bone marrow plasma cells from patients with monoclonal gammopathy of undetermined significance (MGUS) compared to multiple myeloma (MM). Results from this study may identify metabolic differences between pre-malignant and malignant clonal plasma cells in MGUS and MM, respectively. It may also allow researchers better determine the transition from MGUS to MM for the development of potential early diagnostic purposes of preventative strategies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Compare the glutamine anaplerosis activity in bone marrow clonal plasma cells (cPCs) between patients with MGUS and MM using an in vivo and an ex vivo approach.

SECONDARY OBJECTIVES:

I. Compare the tricarboxylic acid (TCA) isotopomer enrichment in the bone marrow plasma obtained from patients with MGUS and MM with the in vivo approach.

II. Determine the peripheral blood enrichment of 13C in the TCA cycle intermediates from patients with MGUS and MM with the in vivo approach.

OUTLINE: Patients are assigned to 1 of 2 groups.

GROUP I (EX-VIVO): After an overnight fast of 6 hours, patients undergo collection of blood samples.

GROUP II (IN VIVO): After an overnight fast of 6 hours, patients receive 13-carbon labeled glutamine or 13-carbon-labeled glucose intravenously (IV) over 90 minutes. Patients also undergo collection of blood and bone marrow aspirate samples.

After completion of study, patient are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* International Myeloma Working Group (IMWG) criteria for the diagnosis of either MGUS or MM

Exclusion Criteria:

* Unable to provide consent
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) > 3
* Hemoglobin < 8 g/dL
* Women who are pregnant
* Prior history of adverse events with conscious sedation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Percent enrichment of 13-Carbon in the tricarboxylic acid (TCA) cycle intermediates within bone marrow plasma cells from patients with monoclonal gammopathy of undetermined significance (MGUS) and multiple myeloma | Up to 1 day
  Will compare the glutamine anaplerosis activity in bone marrow clonal plasma cells between patients with MGUS and multiple myeloma.

SECONDARY OUTCOMES:
Percent enrichment of 13-Carbon in the TCA cycle intermediates within bone marrow plasma from patients with MGUS and multiple myeloma | Up to 1 day
  Will compare the glutamine anaplerosis activity in the plasma cells by assessing the bone marrow plasma between patients with MGUS and multiple myeloma.
Percent enrichment of 13-Carbon in the TCA cycle intermediates within the peripheral blood plasma from patients with MGUS and multiple myeloma | Up to 1 day
  Will compare the peripheral blood enrichment of 13-carbon in the TCA cycle intermediates from patients with MGUS and multiple myeloma.

CONTACTS AND LOCATIONS:
Overall Officials: Wilson I Gonsalves, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Gonsalves WI, Jang JS, Jessen E, Hitosugi T, Evans LA, Jevremovic D, Pettersson XM, Bush AG, Gransee J, Anderson EI, Kumar SK, Nair KS. In vivo assessment of glutamine anaplerosis into the TCA cycle in human pre-malignant and malignant clonal plasma cells. Cancer Metab. 2020 Dec 11;8(1):29. doi: 10.1186/s40170-020-00235-4. PMID 33308307
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials